CLINICAL TRIAL: NCT01860456
Title: Tyrosine Kinase Inhibitors of BCR/ABL: Pharmacokinetic and Pharmacogenetic Study in Patients Affected by Chronic Myeloid Leukemia. Evaluation of Efficacy and Tolerability
Brief Title: TyrosIne Kinase Inhibitors in Chronic Myeloid Leukemia: Efficacy and Tolerability. The TIKlet Study
Acronym: TIKlet
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonello Di Paolo, M.D., Ph.D., Associate Professor of Pharmacology, University of Pisa
Other Study IDs: TIKlet-2012-M1.5
Record Dates: First submitted 2013-05-15; First posted 2013-05-22 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; Imatinib; Nilotinib; Polymorphism, Single Nucleotide; Pharmacokinetics; ATP-Binding Cassette Transporters; SLC Transporters; Treatment outcome; Toxicity
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CML Imatinib/Nilotinib: Patients affected by chronic myeloid leukemia and treated with imatinib or nilotinib
  Interventions: Drug: Imatinib/Nilotinib

INTERVENTIONS:
Drug: Imatinib/Nilotinib — Imatinib: 400 mg/day oral - Nilotinib: 600-800 mg/day oral
  Other Names: Gleevec; Tasigna

SUMMARY:
Rationale

The pharmacokinetics of imatinib and nilotinib, two BCR/Abl tyrosine-kinase inhibitors (TKI), is variable among patients suffering from chronic myeloid leukemia (CML). Transmembrane transporters may play a pivotal role in interindividual variability in TKI disposition. Furthermore, minimum plasma concentrations (Cmin) higher than 1 mg/L could be associated with a higher likelihood of molecular and cytogenetic responses.

The TIKlet study is aimed at evaluating correlations among the pharmacogenetics, pharmacokinetics and treatment efficacy/tolerability of imatinib and nilotinib in CML patients.

1. PATIENTS AND METHODS

1.1. Patients

Patients affected by CML will be enrolled after the informed consent will be signed, according to the following inclusion criteria:

* patients of both sexes,
* age between 18 and 80 years,
* treated with imatinib or nilotinib,
* included in follow-up activities at the participating Hematology Divisions,
* able to give informed consent,
* with a proved compliance with the scheduled treatment.

The administration of other drugs will be allowed, being known the dose and duration of treatment, as well as smoking and herbal products.

Alterations in organ functions or physicochemical exams, body mass index >28 do not represent exclusion criteria.

1.2. Enrollment and follow-up visits

During enrollment visit:

* patients will be informed about the study, their signed informed consent form will be collected and an individual alphanumeric code will be assigned.
* Patients' data will be recorded within the individual case report form (CRF) and a blood sample will be obtained.

At follow-up visits, a blood sample will be collected for therapeutic drug monitoring (TDM) and patients' CRF will be updated.

1.3. Blood samples

After centrifugation, the resulting plasma will be collected for TDM. During the enrollment visit, an aliquot of whole blood will be collected for molecular analyses.

1.4 Laboratory analyses

TDM will be performed by high-performance liquid chromatography systems, then results will be evaluated by a population pharmacokinetic analysis. Single nucleotide polymorphisms will be investigated in the following genes: ABCB1, ABCG2, hOCT1, OCTN1, OATP1A2.

Finally, response to drugs, in terms of Major Molecular Response (MMR) and Complete Cytogenetic Response (CCyR), and tolerability will be evaluated. Any possible correlation among drug disposition, pharmacogenetics and treatment effects will be analyzed.

DETAILED DESCRIPTION:
1. Patients

1.1. Patients

CML patients will be included according to the following inclusion criteria: a) patients of both sexes, b) age between 18 and 80 years, c) treated with imatinib or nilotinib, d) included in the follow-up in the Divisions / Units of Hematology involved in the project e) able to give informed consent to trial participation, f) with a proved compliance with the scheduled treatment.

Patients will be excluded from participation to the study if: a) age <18 or >80 years or b) unable to provide informed consent. The inability to attend the follow-up visits will not be considered an exclusion criterion from the study. In this case, collected data will be used in pharmacokinetic and statistical analyses on the basis of an intention-to-treat criterion.

The following conditions should be noted:

1. the concomitant administration of other drugs will be allowed, provided it will be known the active ingredient, the dose and the period of administration;
2. smoking and herbal products will be allowed but they should be reported on patient's case report form;
3. alterations in liver and kidney functions, body mass index higher than 28, or any other alteration in physicochemical exams do not represent exclusion criteria.

1.2. Sample size

For the purposes of this study it has been estimated that it will need to recruit at least 206 subjects per drug (total, 412 patients), taking into account:

1. the minor allele frequency of the most studied polymorphism evaluated in this research protocol (i.e., 0.3, T allele of the ABCB1 c.3435C>T polymorphism);
2. the 1:1 ratio allele C carriers and patients homozygous for the T allele of the ABCB1 c.3435C>T polymorphism;
3. covariate effects on drug pharmacokinetics will be considered significant when the mean difference in pharmacokinetic parameters will be at least 20%;
4. the power of the study will be 80%;
5. the alpha error will be set at 0.05.

   1.3. Enrollment

   Patient enrollment in the various participating centers will be competitive, up to the achievement of 206 individuals per drug.

   At the first visit, the TIKlet study will be presented to patients who will satisfy the inclusion / exclusion criteria. The following activities will take place:
   * patients will be informed about the characteristics, objectives, and procedures of the study.
   * Consent to study participation will be confirmed by signing the informed consent form.
   * Personal alphanumeric code assignment for patient's identification and privacy.
   * Updating of the enrollment list.
   * Collection of main data of the patient (age, sex, age at diagnosis, clinical chemistry test results as reported in the patient's record and any combination therapies, with their doses and duration) within the individual case report form (CRF).
   * A blood withdrawal (approximately 4 mL) will be performed from a peripheral vein of the forearm. The time at which blood will be withdrawn will be registered within patient's CRF, together with the time elapsed from the last administration of imatinib or nilotinib. For sample handling see section 2.1. "Blood sample handling".
   * The updated list of enrolled patients and individual case report forms will be sent to the Division of Hematology, Dept. of Clinical and Experimental Medicine, University of Pisa

   1.4 Follow-up visits

   According to clinical routine at each participating center, the following activities should be performed during each follow-up visit:
   * Collection of patient's data: clinical chemistry test results, cytogenetic analysis and molecular biology results (BCR/Abl transcript levels), any concomitant therapy, any adverse drug reaction.
   * A blood sample (approximately 4 mL) will be collected from a peripheral vein of the forearm. The time at which blood will be withdrawn will be registered within patient's CRF, together with the time elapsed from the intake of last imatinib or nilotinib dose. For sample handling see section 2.1. "Blood sample handling".

     2. Laboratory analyses

   Laboratory analyses will be conducted at the Division of Pharmacology, Department of Clinical and Experimental Medicine, University of Pisa (measurement of drug plasma concentrations, pharmacogenetic analyses) and at the Department of Pharmacology, University of Bologna (pharmacogenetic analyses).

   2.1. Blood sample handling

   Each tube containing the patient's whole blood, plasma or DNA (see below) and used for the execution of therapeutic monitoring or pharmacogenetic analyses will be identified by a) the patient's code and b) the date of execution of blood withdrawal.

   All blood samples will be collected in lithium-heparin Vacutainer® tubes, then they will be stored at 4 °C until centrifugation. The sample will be centrifuged and the resulting plasma (1.5 mL) will be collected and stored in a tube for therapeutic drug monitoring. Only during the enrollment visit, an aliquot of whole blood (0.5 mL) will be collected in a sterile eppendorf for molecular analyses. Both samples will be stored at -20 °C for a maximum of 2 weeks, then they will be sent to the Dept. of Clinical and Experimental Medicine, University of Pisa.

   For sample storage see section 2.7. "Biological sample storage".

   2.2 Measurement of plasma concentration of drugs

   The measurement of plasma concentrations of imatinib and its active metabolite, and nilotinib will be conducted by a high-performance liquid chromatography (HPLC) method using commercially available kits (Chromsystems GmbH, Munich, Germany) on Waters Breeze and Alliance instruments (Waters, USA).

   Briefly, solid-phase extraction columns will be balanced with Equilibration buffers 1 and 2, then the internal standard and plasma (0.5 mL) will be added. The column will be centrifuged, and subsequently washed with Wash buffer and water for HPLC. The eluate will be collected by centrifugation, diluted with water for HPLC and injected (0.025 mL) into the HPLC system for the execution of the analysis. The peak area of the analytes of interest (imatinib and its active metabolite, nilotinib and internal standard) will be recorded and the actual concentration of drug in plasma will be obtained by comparison with standard calibration curves for each day of analysis.

   The HPLC analyses will be carried out on a weekly basis. The reports of the analysis will be sent to the Divisions / Units of Hematology and registered into both the patient's medical record and study CRFs.

   2.3. Pharmacokinetic analyses

   Plasma concentrations of imatinib/active metabolite and nilotinib will be analyzed trough a population pharmacokinetic analysis according to a nonlinear mixed-effects modeling approach, using the NONMEM software, version 7.2. The Xpose and PsN packages will be used to check database, for model diagnostic and covariate testing. Former models for imatinib/metabolite and nilotinib will be 1- and 2-compartment models with first-order elimination and parameterized in terms of apparent drug clearance (CL/F), volume of distribution (V/F) and absorption constant (ka), while the residual error will be modeled as additive, proportional or mixed (additive and proportional) error. The availability of records, goodness-of-fit plots and the precision of parameter estimates, together with a generalized additive modeling procedure (GAM) implemented in the Xpose package, will be adopted for model development and to explore correlations among the covariates. In particular, age, weight, body mass index, liver (ALT, AST) and renal function (creatinine plasma concentration), albumin and α1-acid glycoprotein plasma concentrations and results of pharmacogenetic analyses will be considered as possible covariates. A stepwise covariate model building will be performed with forward inclusion and backward exclusion. In particular, a decrease in the objective function value (OFV) greater than 3.84 points (i.e., p<0.05) and 6.63 points (i.e., p<0.01) will be the criteria used in the forward inclusion and backward exclusion steps, respectively. The goodness of the final model will be checked by bootstrap analysis using the PsN and Xpose packages and calculating η-shrinkage. The area under the plasma concentration-time curve from time zero up to infinity (AUC) and terminal elimination half-life (t1/2) will be calculated from the individual empirical Bayes estimates (EBE) from the final population pharmacokinetic model as follows:

   AUC=(Total daily dose)/(CL/F) t1/2=ln(2)/kel where kel is imatinib elimination constant.

   2.4. Pharmacogenetic analyses

   The aliquot of frozen whole blood will be employed for the extraction of genomic DNA with a suitable kit (Qiagen, Milan, Italy) following manufacturer's instructions and the nucleic acid will be stored at -80 ° C until the time of analysis in sterile tube bearing the identification code of the patient.

   Single nucleotide polymorphisms (SNPs) of the following genes will be assayed: ABCB1, ABCG2, hOCT1, OCTN1, OATP1A2. SNPs will be evaluated by specific kits from Applied Biosystems (Life Sciences, Milan, Italy) on an ABI Prism 7900HT Sequence Detection System (Life Sciences). Each analysis will be performed in triplicate. Genotypes will be automatically identified through the software SDS (Life Sciences). Frequency of alleles and genotypes according to the Hardy-Weinberg law, haplotype and linkage disequilibrium analysis will be performed using Arlequin software package.

   2.5. Treatment effectiveness and tolerability

   The response to the therapy with imatinib will be evaluated in agreement with criteria recently published and adopted. In particular, results from chemical, biochemical and molecular analyses will be performed every 2 weeks during the first 3 months of treatment, then cytogenetic (metaphase chromosomal banding assay) and molecular analyses (quantification of BCR-ABL transcription levels in plasma by real-time-PCR) were performed every 6 and 3 months, respectively, until the attainment of a complete response. The time to complete cytogenetic response (CCyR) and to major molecular response (MMR) will be defined as the length of time elapsed from diagnosis and response attainment for every patient.

   Furthermore, treatment-associated adverse reactions (i.e., nausea and vomiting, periorbital oedema, cramps and myalgia, neutropenia, skin and liver toxicities) will be identified and scored according to the Common Toxicity Criteria-NCI grading system (version 3).

   2.6. Statistical analysis

   The results will be analyzed in aggregate form. Parameter of dispersion (standard deviation, range), central indexes (mean, median) and distribution (i.e., Kolmogorov-Smirnov test) will be calculated. The most appropriate statistical tests (ANOVA, Fisher test, etc.) will be applied to investigate any possible difference between groups, and the level of significance will be set at p = 0.05. The identification of cut-off values for parameters predictive of efficacy / tolerability (plasma concentrations, polymorphisms) will be pursued trough ad hoc analyses (receiver operating characteristics analysis, evaluation of positive and negative predictive values).

   2.7. Biological sample storage

   All biological samples [whole blood (0.5 mL), plasma (1.5 mL) and genomic DNA] will be stored at the Division of Pharmacology, Department of Clinical and Experimental Medicine, University of Pisa. Aliquots of DNA samples for pharmacogenetic analyses will be stored at the Department of Pharmacology, University of Bologna.

   Each sample will be identified by the individual alphanumeric code assigned to every patient. According to protocol, patients may require the destruction of their own biological samples.

   2.8. Authorship

   The criteria declared by the ICMJE (International Committee of Medical Journal Editors) will be adopted for authorship definition.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by chronic myeloid leukemia
* Age limits: 18-80 years
* Male and female patients
* Treatment with imatinib/nilotinib since at least 3 weeks
* Optimal adherence
* Signed informed consent

Exclusion Criteria:

* Age <18 or >80 years
* Poor adherence
* Inability to attend follow-up visits
* Lack of signed informed consent

Concomitant administration of other drugs will be allowed, but active pharmacological agents, their dose and duration of treatment should be recorded.

Smoking is not considered an exclusion criterium, but it should be noticed and recorded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by CML from Hematology Units
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage differences in Imatinib/Nilotinib pharmacokinetic parameters according to Solute Carrier (SLC) and ATB-Binding Cassette (ABC) transporters polymorphisms in chronic myeloid leukemia patients | 2 years
  Percentage difference in drugs pharmacokinetic parameters (apparent clearance [CL/F], minimum plasma concentration at steady state [Cmin,ss], area under the time concentration curve [AUC], terminal elimination half-life [t1/2]) according to polymorphisms of SLC and ABC transporters (wild-type homozygous vs. heterozygous and polymorphic homozygous patients)

SECONDARY OUTCOMES:
Time to Complete Cytogenetic Response (Time-to-CCyR) and Major Molecular Response (Time-to-MMR) | 2 years
  The time-to-CCyR and the time-to-MMR will be the time elapsed from diagnosis and response attainment on the basis of metaphase chromosomal banding assay and BCR-ABL transcriptional plasma level quantification by real-time-PCR, respectively
Time-to-CCyR or Time-to-MMR and Cmin,ss values or SLC / ABC genotype | 2 years
  The time to attain optimal response to drugs in terms of CCyR or MMR according to Cmin,ss values (<1 mg/L or >1 mg/L) and SLC / ABC genotypes (wild-type homozygous vs. heterozygous and polymorphic homozygous)
Percentage of patients who achieve MMR/CCyR and Cmin,ss values or SLC/ABC genotype | 2 years
  The percentage of patients who achieve MMR/CCyR according to Cmin,ss values (<1 mg/L or >1 mg/L) and SLC / ABC genotypes (wild-type homozygous vs. heterozygous and polymorphic homozygous)
Number of patients with Adverse Drug Reactions and Cmin,ss values or SLC / ABC genotype | 2 years
  Number of patients with Adverse Drug Reactions according to Cmin,ss values (<1 mg/L or >1 mg/L) and SLC / ABC genotypes (wild-type homozygous vs. heterozygous and polymorphic homozygous)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Galimberti, MD, PhD, Principal Investigator — Department of Clinical and Experimental Medicine, University of Pisa; Antonello Di Paolo, MD, PhD, Principal Investigator — Department of Clinical and Experimental Medicine, University of Pisa
Locations (2):
- Italy (2):
  - Unit of Hematology, Azienda Ospedaliero Universitaria Pisana, Pisa
  - Division of Hematology and Transplants, University of Siena, Siena

REFERENCES:
- [Result] Di Paolo A, Polillo M, Capecchi M, Cervetti G, Barate C, Angelini S, Guerrini F, Fontanelli G, Arici R, Ciabatti E, Grassi S, Bocci G, Hrelia P, Danesi R, Petrini M, Galimberti S. The c.480C>G polymorphism of hOCT1 influences imatinib clearance in patients affected by chronic myeloid leukemia. Pharmacogenomics J. 2014 Aug;14(4):328-35. doi: 10.1038/tpj.2014.7. Epub 2014 Mar 4. PMID 24589908
- [Result] Carulli G, Barate C, Marini A, Ottaviano V, Cervetti G, Fontanelli G, Guerrini F, Arici R, Guerri V, Di Paolo A, Polillo M, Ferreri MI, Galimberti S, Petrini M. Reduced circulating B-lymphocytes and altered B-cell compartments in patients suffering from chronic myeloid leukaemia undergoing therapy with Imatinib. Hematol Oncol. 2015 Dec;33(4):250-2. doi: 10.1002/hon.2156. Epub 2014 Sep 25. No abstract available. PMID 25256816
- [Result] Crea F, Di Paolo A, Liu HH, Polillo M, Clermont PL, Guerrini F, Ciabatti E, Ricci F, Barate C, Fontanelli G, Barsotti S, Morganti R, Danesi R, Wang Y, Petrini M, Galimberti S, Helgason CD. Polycomb genes are associated with response to imatinib in chronic myeloid leukemia. Epigenomics. 2015 Aug;7(5):757-65. doi: 10.2217/epi.15.35. Epub 2015 Sep 7. PMID 26343356
- [Result] Galeotti L, Ceccherini F, Domingo D, Laurino M, Polillo M, Di Paolo A, Barate C, Fava C, D'Avolio A, Cervetti G, Guerrini F, Fontanelli G, Ciabatti E, Grassi S, Arrigoni E, Danesi R, Petrini M, Cornolti F, Saglio G, Galimberti S. Association of the hOCT1/ABCB1 genotype with efficacy and tolerability of imatinib in patients affected by chronic myeloid leukemia. Cancer Chemother Pharmacol. 2017 Apr;79(4):767-773. doi: 10.1007/s00280-017-3271-3. Epub 2017 Mar 13. PMID 28289867
- [Result] Galimberti S, Bucelli C, Arrigoni E, Barate C, Grassi S, Ricci F, Guerrini F, Ciabatti E, Fava C, D'Avolio A, Fontanelli G, Cambrin GR, Isidori A, Loscocco F, Caocci G, Greco M, Bocchia M, Aprile L, Gozzini A, Scappini B, Cattaneo D, Scortechini AR, La Nasa G, Bosi A, Leoni P, Danesi R, Saglio G, Visani G, Cortelezzi A, Petrini M, Iurlo A, Di Paolo A. The hOCT1 and ABCB1 polymorphisms do not influence the pharmacodynamics of nilotinib in chronic myeloid leukemia. Oncotarget. 2017 Sep 30;8(50):88021-88033. doi: 10.18632/oncotarget.21406. eCollection 2017 Oct 20. PMID 29152138
- [Result] Galimberti S, Grassi S, Barate C, Guerrini F, Ciabatti E, Perutelli F, Ricci F, Del Genio G, Montali M, Barachini S, Giuliani C, Ferreri MI, Valetto A, Abruzzese E, Ippolito C, Iurlo A, Bocchia M, Sicuranza A, Martino B, Iovino L, Buda G, Salehzadeh S, Petrini M, Di Paolo A, Mattii L. The Polycomb BMI1 Protein Is Co-expressed With CD26+ in Leukemic Stem Cells of Chronic Myeloid Leukemia. Front Oncol. 2018 Dec 6;8:555. doi: 10.3389/fonc.2018.00555. eCollection 2018. PMID 30574454
- [Result] Abruzzese E, Aureli S, Bondanini F, Ciccarone M, Cortis E, Di Paolo A, Fabiani C, Galimberti S, Malagola M, Malato A, Martino B, Trawinska MM, Russo D, de Fabritiis P. Chronic Myeloid Leukemia and Pregnancy: When Dreams Meet Reality. State of the Art, Management and Outcome of 41 Cases, Nilotinib Placental Transfer. J Clin Med. 2022 Mar 24;11(7):1801. doi: 10.3390/jcm11071801. PMID 35407407